CLINICAL TRIAL: NCT06925672
Title: Assessment Of Knowledge, Attitude and Perception of Pregnant Women Regarding Medications Use
Brief Title: Knowledge, Attitude and Perception of Pregnant Women Regarding Medications
Status: Active, not recruiting | Type: Observational
Sponsor: Rania Hassan Mostafa (Other)
Responsible Party: Sponsor-Investigator, Rania Hassan Mostafa, Associate Professor, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: FMASU MS 185/2025
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Medications in Pregnancy
Keywords: pregnancy; medication; attitude; perception; knowledge; teratogenic
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women attending the Ain shams University Maternity Hospital
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — This is an anonymous questionnaire; based upon previous similar studies.
  The questionnaire comprises closed-ended questions categorized into four sections, along with fifth section consisting of statements pertaining to respondents' beliefs:
  A. Section A (10 items) will contain information about the participant's socio-demographic and health related characteristics.
  B. Section B (7 items) will assess their knowledge about medication use and restriction, during pregnancy.
  C. Section C (4 items) will assess their attitude about medication. D. Section D (4 items) will assess the source of their information. E. Section E (9 statements) will assess their beliefs about medications use during pregnancy.
  This questionnaire will be presented in its Arabic version.
  Other Names: survey

SUMMARY:
The goal of this observational study is to learn about the pregnant women's knowledge, attitude, and perception regarding the use of medications in pregnancy. The main question it aims to answer is:

What is the present knowledge, attitude, and perception of pregnant women regarding medication use?

Participants (pregnant women) already attending the antenatal clinic for routine follow-up will answer survey questions about their knowledge, attitude, and beliefs about medication use and restriction during pregnancy, as well as the source of their information.

DETAILED DESCRIPTION:
This is a descriptive cross-sectional study (survey) that will be held at Ain shams University Maternity Hospital.

The protocol approval will be sought from the ethical committee of department of Obstetrics and Gynecology, Ain Shams University.

• Data collection (the questionnaire): The study will use anonymous questionnaire; based upon previous similar studies.

The questionnaire comprises closed-ended questions categorized into four sections, along with fifth section consisting of statements pertaining to respondents' beliefs:

A. Section A (10 items) will contain information about the participant's socio-demographic and health related characteristics.

B. Section B (7 items) will assess their knowledge about medication use and restriction, during pregnancy.

C. Section C (4 items) will assess their attitude about medication. D. Section D (4 items) will assess the source of their information. E. Section E (9 statements) will assess their beliefs about medications use during pregnancy.

This questionnaire will be presented in its Arabic version and pre-tested on 15 pregnant women to evaluate the construct and content validity, as well as to determine if any modifications to wording are necessary. These participants will not be included in the final analysis.

The questionnaire will be distributed to pregnant women who attend the hospital for their routine antenatal check-up visits. In instances where women are unable to read or write, the principal investigator and attending house officer in the unit will provide assistance in reading and explaining the questions to facilitate the completion of the questionnaire.

* Data will be collected and recorded.
* Statistical analysis will be done accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending the Ain shams University Maternity Hospital

Exclusion Criteria:

* Pregnant ladies refusing to participate in study.
* Pregnant ladies needing immediate transport to emergency department.
* Pregnant ladies needing immediate intervention.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who attend the Ain shams University Maternity Hospital for their routine antenatal check-up visits
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge of pregnant women regarding medication use and restriction in pregnancy. | Once at recruitment
  Degree of knowledge (information) that the pregnant women have about medication use and restriction during pregnancy, as well as the source of their information, as assessed by answering the questions in sections B and D in the questionnaire.

SECONDARY OUTCOMES:
Attitude of pregnant women regarding medication use | Once at recruitment
  The attitudes of the pregnant women towards medication use during pregnancy, as assessed by answering the questions in section C in the questionnaire.
Perception and beliefs of pregnant women regarding medication use and restriction | Once at recruitment
  The beliefs of the pregnant women regarding medication use during pregnancy, as assessed by answering the questions in section E in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khairy, MD, Study Chair — Faculty of Medicine, Ain Shams University.; Ebtihal M Eltaieb, MD, Study Director — Faculty of Medicine, Ain Shams University.
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, the questionnaire used, and the analytic code will be made available on OSF platform.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The study protocol and the questionnaire used will be available starting (May 2025) till (May 2030) The analytic code will be available after publishing the results (expected by May 2026) for 5 years
Access Criteria: The study protocol, the questionnaire used, and the analytic code will be made PUBLICLY available on OSF platform.
URL: https://osf.io/